CLINICAL TRIAL: NCT01985204
Title: Assessment of the Improvement of the Cardiovascular Risk Profile in Obese Women After Correction of Iodine Deficiency
Brief Title: Iodine Supplementation in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Isabelle Aeberli, PhD, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK 2013-N-24
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Iodine Deficiency; Subclinical Hypothyroidism
Keywords: iodine; thyroid hormones; obesity; TSH; dyslipidemia; insulin resistance
MeSH Terms: conditions — Obesity; Dyslipidemias; Insulin Resistance | interventions — Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Dietary Supplement: Placebo tablet
- Intervention (Experimental): Iodine tablet
  Interventions: Dietary Supplement: Iodine tablet

INTERVENTIONS:
Dietary Supplement: Iodine tablet — Iodine tablets containing 200 ug iodine as potassium iodate
  Arms: Intervention
Dietary Supplement: Placebo tablet — Placebo tablet without iodine
  Arms: Placebo

SUMMARY:
The study hypothesis is that iodine supplementation will lower serum TSH and leptin concentrations and thereby improve the lipid and glucose profile.

DETAILED DESCRIPTION:
The study will be a double blind, placebo controlled intervention study in obese women living in the Atlas foot mountains in Morocco, an iodine deficient area. Eligible subjects will be randomized into intervention and control group and will receive the respective supplement for 6 months. At baseline, midpoint and endpoint anthropometric as well as metabolic profile will be assessed. A health questionnaire will further be administered monthly when the tablets for the following month are distributed. Urine samples to determine iodine status will also be collected monthly.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (20 to 50 years)
* Body mass index 27 to 40 kg/m2
* Having received oral and written information about the aims and procedures of the study
* Willing to comply with the study procedure
* Having provided oral and written informed consent

Exclusion Criteria:

* Chronic disease or gastrointestinal disorders
* Nodular goiter
* Regular use of medication (except oral contraceptives)
* Pregnancy or lactation
* Subject who cannot be expected to comply with study protocol

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in TSH (thyroid-stimulating hormone) | change from baseline to 6 months
change in fasting insulin | change from baseline to 6 months
change in the LDL cholesterol/ HDL cholesterol ratio | change from baseline to 6 months

SECONDARY OUTCOMES:
fasting glucose | baseline, 3 months and 6 months
plasma leptin | baseline, 3 months and 6 months
LDL cholesterol | baseline, 3 months and 6 months
HDL cholesterol | baseline, 3 months and 6 months
Urinary iodine | change from baseline to 6 months

OTHER OUTCOMES:
T3 | baseline, 3 months and 6 months
T4 | baseline, 3 months and 6 months
total cholesterol | baseline, 3 months and 6 months
TSH | 3 months
leptin | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Aeberli, PhD, Principal Investigator — ETH Zurich (Switzerland)
Locations (2):
- Morocco (2):
  - Universite Caddi Ayad, Faculte de Medecine et de Pharmacie, Marrakesh
  - University Cadi Ayyad, Faculte des Sciences, Marrakesh

REFERENCES:
- [Derived] Herter-Aeberli I, Cherkaoui M, El Ansari N, Rohner R, Stinca S, Chabaa L, von Eckardstein A, Aboussad A, Zimmermann MB. Iodine Supplementation Decreases Hypercholesterolemia in Iodine-Deficient, Overweight Women: A Randomized Controlled Trial. J Nutr. 2015 Sep;145(9):2067-75. doi: 10.3945/jn.115.213439. Epub 2015 Jul 22. PMID 26203098